CLINICAL TRIAL: NCT02225912
Title: A Study to Evaluate the Efficacy of the Nasal Antiseptic, PrevinC, When Administered for the RiskReduction of Rhinitis in Subjects Who Work for Child Day Care Centers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BioHealth Technologies Inc. (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Triple
Other Study IDs: Previn-C
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2014-08

CONDITIONS: Upper Respiratory Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- PrevinC (Experimental): PrevinC contains isopropyl alcohol, sesame oil, aloe vera oil extract, and lemon oil.
  Interventions: Other: PrevinC
- Control solution (Placebo Comparator): The control solution (distilled water and lemon oil) was similar in color, oily consistency and odor to that of PrevinC.
  Interventions: Drug: placebo

INTERVENTIONS:
Other: PrevinC
  Arms: PrevinC
Drug: placebo
  Arms: Control solution

SUMMARY:
The hypothesis was to establish whether the use of PrevinC administered nasally 2-3 times a day will prevent upper respiratory infections in otherwise healthy adults working in child day care centers.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide written informed consent prior to the conduct of any study
* Male or female
* 18-65 years of age
* Inclusive
* Employed by one of seven selected Day Care Centers

Exclusion Criteria:

* Recent symptoms of upper respiratory infection, respiratory disease
* Received medication for colds or allergies within 3 weeks of enrolling
* Had nasal surgery within 2 months of enrolling
* Had a pierced nose or wore nose jewelry

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Rhinitis | weekly from February 2005 to May 2005, up to 3 months
  The incidence of rhinitis was measured on a weekly basis through evaluation of study diaries.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sunflower Preschool & Day Care, Hialeah, Florida
  - Sunflower Preschool Childcare, Miami, Florida
  - Sunflowers Academy, Miami, Florida
  - Sunflowers Preschool Childcare, Miami, Florida
  - Mt Sinai Day Care, Miami Beach, Florida